CLINICAL TRIAL: NCT03452410
Title: Positive Diagnosis of Vestibular Neuritis Using Fluid Attenuated Inversion Recuperation (FLAIR) Sequence, One Hour After Intravenous Gadolinium Injection, on a 1.5 Tesla
Brief Title: MRIPositive Diagnosis of Vestibular Neuritis Using Fluid Attenuated Inversion Recuperation (FLAIR) Sequence on a 1.5 Tesla
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6786
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2018-02

CONDITIONS: Vestibular Neuritis
Keywords: Vestibular neuritis; Magnetic resonance imaging (MRI); Vertigo; Fluid attenuated inversion recuperation (FLAIR)
MeSH Terms: conditions — Vestibular Neuronitis; Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our objective is to allow positive MRI diagnosis of vestibular neuritis by highlighting contrast enhancement of the vestibular nerve on the pathological side of the FLAIR sequence acquired 1h after intravenous gadolinium injection in patients with typical vestibular neuritis. At present, the diagnosis is based on a combination clinical examination / video-head impulse test, and no imaging examination allows the diagnosis to be positive.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Presence of a typical unilateral vestibular neuritis during the ENT examination with videonystagmography
* Subject having his agreement for the use of his medical data for research purposes.

Exclusion Criteria:

* Special clinical forms of the disease: doubtful or atypical forms, especially the presence of deafness
* Treatments and related interfering diseases, antecedents: antecedents of neuritis for controls, presence of vertigo, bilateral involvement
* Impossibility to give the subject information enlightened (subject in emergency situation, difficulties of understanding the subject, ...)
* Subject under the protection of justice
* Subject under guardianship or curatorship

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with typical unilateral vestibular neuritis during ENT examination with videonystagmograph
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-02-23 (Actual); Study Completion 2019-02-23 (Actual)

PRIMARY OUTCOMES:
Diagnosis of vestibular neuritis | one hour after intravenous gadolinium injection

CONTACTS AND LOCATIONS:
Locations (1):
- Service Imagerie 1, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No